CLINICAL TRIAL: NCT04415814
Title: Unilateral Versus Bilateral Pedicle Screw Fixation for Lumbar Degenerative Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1123
Record Dates: First submitted 2020-05-23; First posted 2020-06-04 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-04

CONDITIONS: Fusion of Spine
Keywords: degenerative spine; unilateral fixation of the spine; fusion of the lumbar spine; posterior stabilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Unilateral Pedicle Screw Fixation) (Experimental): Patients will undergo stabilizing surgery on the lumbar spine for degenerative diseases of the spine. Pedicular screws will be installed unilaterally, which means on one side of the spinous processes. The system will be fixed with standard rod and blockers.
  Interventions: Procedure: Unilateral Pedicle Screw Fixation
- Group 2 (Bilateral Pedicle Screw Fixation) (Active Comparator): Patients will undergo stabilizing surgery on the lumbar spine for degenerative diseases of the spine. Pedicular screws will be installed bilaterally, which means on the both sides of the spinous processes. The system will be fixed with standard rods and blockers.
  Interventions: Procedure: Bilateral Pedicle Screw Fixation

INTERVENTIONS:
Procedure: Unilateral Pedicle Screw Fixation — Pedicle screws are installed unilaterally on the one side of the vertebrae and fixed with rod
  Arms: Group 1 (Unilateral Pedicle Screw Fixation)
Procedure: Bilateral Pedicle Screw Fixation — Pedicle screws are installed bilaterally on the both sides of the vertebrae and fixed with rods
  Arms: Group 2 (Bilateral Pedicle Screw Fixation)

SUMMARY:
Determining the treatment strategy for patients with degenerative diseases of the spine is extremely difficult, without an accurate understanding of the nature of stress distribution in the vertebral-motor segments of the spine, as well as biomechanical changes that are associated with degenerative diseases of the spine. In this clinical study, we want to compare the use of unilateral and bilateral transpedicular fixation for treating the patients with degenerative diseases of the lumbar spine.

DETAILED DESCRIPTION:
It is planned to use posterior stabilization without interbody fusion. In the postoperative period, all the patients receive antibacterial and analgesic therapy. The early postoperative period is spent in a hospital. Repeated appearances for control examinations (3, 6, 12 months) are provided for physical examination (EQ-5D, Oswestry Disability Index) and performing radiographs or computed tomography (CT) of the spine. All patients undergo a standard rehabilitation course.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient to participate in the study;
* Patients with degenerative diseases of the lumbar spine.
* The opportunity for observation during the entire study period (12 months);
* Mental adequacy, ability, willingness to cooperate and follow the doctor's recommendations.

Exclusion Criteria:

* The refusal of a patient from surgery
* The presence of contraindications to surgery
* Severe forms of diabetes (glycosylated hemoglobin >9%);
* Blood diseases (thrombopenia, thrombocytopenia, anemia with Hb< 90g\l);
* The unwillingness of the patient to conscious cooperation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
fusion rate of the operated spine segment | in 3 months after surgery
  Control CT/Radiography examination
fusion rate of the operated spine segment | in 6 months after surgery
  Control CT/Radiography examination
fusion rate of the operated spine segment | in 12 months after surgery
  Control CT/Radiography examination

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Lychagin, MD, PhD, Study Chair — IM Sechenov University
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No